CLINICAL TRIAL: NCT00141635
Title: Enhancing the Status of Quality of Life Diagnostics in Caring for Breast Cancer Patients: Results From a Multilevel Implementation Study in a Regional Tumor Centre
Brief Title: Implementation of Quality of Life Diagnostics and Therapy
Status: Completed | Type: Observational
Sponsor: Tumor Center Regensburg (Other)
Other Study IDs: TUZ-QL-IP-03; 3.5/8203-1/117/02
Record Dates: First submitted 2005-08-31; First posted 2005-09-01 (Estimated); Last update posted 2005-09-01 (Estimated); Status verified 2005-08

CONDITIONS: Breast Neoplasms
Keywords: Quality of Life; Breast Cancer; Referee's Report; Diagnostics; Therapy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

INTERVENTIONS:
Behavioral: physio,pain,psychotherapy;social,nutrit.counselling&sports

SUMMARY:
Implementation and Evaluation of Implementation of Quality of Life Diagnostics and Therapy in Individual Patients with Breast Cancer. A prospective study including 170 patients, 5 clinics and 38 general practitioners as coordinating doctors for quality of life therapies. Correlational study including several comparisons such as patients and their doctors.

DETAILED DESCRIPTION:
Improving cancer patients' quality of life (QL) requires that QL-diagnostics, the availability of QL-enhancing treatment options and treatment decisions are being integrated into a clinical path. This description presents the development and implementation of such a clinical path in the Tumorcenter Regensburg.

The acting persons and institutions in this clinical path are the breast cancer patients, the hospitals, the family doctors or gynaecologists, and a QL-study team. Starting point is the QL-assessment either in the hospital or in doctors' practice (EORTC QLQ-C30 plus BR-23). The caring physician documents the patients' health status. Based on these two pieces of information, the QL-study team writes up a medical/QL-opinion plus therapy recommendation. This report is sent to the caring physician. The effectiveness of the therapy recommendation is assessed in the following QL-assessment. This clinical path is implemented via three interrelated methods of implementation: local opinion leaders, outreach visits, and quality circle.

A total of 38 physicians were made familiar with QL-diagnostics through outreach visits, and 12 opinion leaders were identified and convinced to support this project. The quality circle provided regular CME meetings on QL-enhancing therapy options (pain control, psychotherapy, physiotherapy, nutrition, social rehabilitation). A total of 170 QL-reports were sent to physicians. All 38 doctors found the QL-profiles comprehensible and the therapy recommendations clinically relevant. The most common QL-problems were emotional functioning, fatigue, and arm/shoulder problems.

QL-diagnostics is a new way to individualise and to rationalise patient care. It transforms the QL-concept into a decision-relevant, integral part of a clinical path that aims to provide high quality patient care.

ELIGIBILITY:
Inclusion Criteria:

* All patients with primary breast cancer in the county of Regensburg, Amberg and Sulzbach-Rosenberg in the year 2003 to June 2004 submitted by coordinating physicians who were trained in quality of life questionnaires and profiles.

Exclusion Criteria:

* Secondary breast cancer, patients who refused to participate, patients incapable of filling out questionnaires, male patients, pregnant patients, age below 18 yrs.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190
Dates: Start 2002-12; Study Completion 2004-06

CONTACTS AND LOCATIONS:
Overall Officials: Monika KS Klinkhammer-Schalke, MD, Study Chair — Tumor Center Regensburg; Michael MK Koller, Ph.D., Principal Investigator — University of Marburg, Institut of Theoretical Surgery; Brigitte BE Ernst, MD, Principal Investigator — General Practitioner, Bad Abbach; Ferdinand FH Hofstädter, MD, Prof., Principal Investigator — Tumor Center Regensburg; Wilfried WL Lorenz, MD, Prof., Principal Investigator — Tumor Center Regensburg
Locations (1):
- Tumorzentrum Regensburg, Regensburg, Bavaria, Germany

REFERENCES:
- [Background] Koller M, Lorenz W. Quality of life: a deconstruction for clinicians. J R Soc Med. 2002 Oct;95(10):481-8. doi: 10.1177/014107680209501002. No abstract available. PMID 12356967
- See also: Related Info — http://www.tumorzentrum-regensburg.de